CLINICAL TRIAL: NCT06590038
Title: Psychotherapy Feasibility and Acceptability Pilot of the Carolina Recovery From Depression Protocol (CARED): A Novel Rapid Treatment Paradigm for Depression
Brief Title: Psychotherapy Feasibility Pilot of the Carolina Recovery From Depression Protocol
Acronym: CARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The Foundation of Hope for Research and Treatment of Mental Illness (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-1988
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Depression, Unipolar
Keywords: Depression; Major Depressive Disorder; Psychotherapy; Single Session Intervention
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy Arm (Experimental)
  Interventions: Behavioral: Single Session Psychotherapy Intervention

INTERVENTIONS:
Behavioral: Single Session Psychotherapy Intervention — This is a single session intervention which incorporates elements from second- and third wave psychotherapies (Acceptance and Commitment Therapy and Behavioral Activation), as well as basic psychoeducation. Session will take approximately three hours in total, with the option for breaks between blocks of session.

SUMMARY:
The goal of this clinical trial is to learn whether an single session intervention can reduce psychological impairment in adult individuals with moderate depression. The main questions it aims to answer are:

Is this evidence-based intervention acceptable to study participants? Is this evidence-based intervention feasible to implement in a single session? Is there evidence that the evidence-based intervention reduces psychological impairment in adults with moderate to severe depression?

Participants will complete:

* an in-depth diagnostic screening interview prior to enrollment
* a set of mental health questionnaires at baseline and two weeks post-intervention
* a 3-hour, evidence-based, single session psychotherapeutic intervention with a trained clinician

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Able to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study
* Speak and understand English
* Diagnostic and Statistical Manual (DSM)-5 diagnosis of major depressive disorder (MDD) as confirmed by semi-structured clinical assessment
* Meet a cutoff of at least a moderate depression score on the Beck Depression Inventory (BDI-II) (≥ 20)

Exclusion Criteria:

* Participants must not have current active suicide intent as determined by the Columbia Suicide Severity Rating Scale (C-SSRS)
* Participants must not meet criteria for current severe substance use disorder, anorexia nervosa, or active psychosis as assessed by psychodiagnostic assessment
* Any participants taking psychotropic medication must be on a stable dose for at least 4 weeks with no planned dose changes within the next 4 weeks.
* Participants able to birth must not be pregnant or breastfeeding.
* Participants may not have any medical or neurological illness for which symptom presentation or treatment could interfere with study participation
* Participants may not have undergone prior brain surgery
* Participants may not have any brain devices/implants, including cochlear implants and aneurysm clips
* Participants may not have had brain injury or concussion within the last three months
* Participants may not have a history of brain injury requiring current treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
CARED Treatment Experience Survey | Immediately post-intervention (same day)
  A brief survey which probes the qualitative experience of participants during the intervention (i.e., tolerability, their level of engagement, satisfaction with treatment). Participants respond to eight items, rated on a 4-point Likert scale (1 - Not at all to 4 - Completely) to indicate their level of agreement with each item. Higher scores on the measure indicate greater tolerability, satisfaction, and endorsement of treatment. Total possible scores range from 8 to 32.

SECONDARY OUTCOMES:
Change from baseline on Behavioral Activation Scale at two weeks post-intervention | Baseline and Two Weeks post-intervention
  The Behavioral Activation Scale is a measure which assesses participant current levels of behavioral activation in the context of current depression. Participants respond to twenty-five items, rated on a 7-point Likert scale (0 - Not at all to 6 - Completely) to indicate their activation levels during the past week. Higher scores on the measure indicate greater activation (i.e., higher functioning) and lower scales indicate lower activation. Total possible scores range from 0 to 150.
Change in baseline Repetitive Thinking Questionnaire - 10 item form to two weeks post-intervention | Baseline and Two weeks post-intervention
  The Repetitive Thinking Questionnaire- 10 item form is a well-validated measure that assesses trait-like repetitive negative thinking (e.g., worry, cognitive rumination) during times of distress. Participants respond to ten items, rated on a 5-point Likert scale (1 - Not true at all to 5 - Very True) to indicate to what extent they agree with each statement. Higher scores on the measure indicate greater trait engagement in repetitive negative thinking. Total possible scores range from 10 to 50.
Change from baseline on Snaith-Hamilton Pleasure Scale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Snaith-Hamilton Pleasure Scale is a measure which assesses participant capacity to experience pleasure in the past few days. Participants respond to fourteen items, rated on a 4-point Likert scale (0 - Strongly disagree to 4 - Strongly agree) to indicate their hedonic capacity over the last few days. Higher scores on the measure indicate greater hedonic capacity, or capacity to experience pleasure. Total possible scores range from 0 to 56.
Change from baseline on Behavioral Inhibition and Behavioral Activation Scale - Inhibition Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Behavioral Inhibition and Behavioral Activation Scale- Inhibition subscale is a well-validated measure that assesses for trait-like behavioral inhibition, similar to overcontrol. Participants respond to seven items, rated on a 4-point Likert scale (1 - Very true for me to 4 - Very false for me) to indicate their general behavioral inhibition. Higher scores on the measure indicate higher inhibition. Total possible scores range from 7 to 28.
Change from baseline on Behavioral Inhibition and Behavioral Activation Scale - Activation Drive Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Behavioral Inhibition and Behavioral Activation Scale- Activation Drive subscale is a well-validated measure that assesses for trait-like behavioral drive, similar to goal seeking activation. Participants respond to four items, rated on a 4-point Likert scale (1 - Very true for me to 4 - Very false for me) to indicate their general behavioral drive. Higher scores on the measure indicate higher drive/goal seeking. Total possible scores range from 4 to 16.
Change from baseline on Behavioral Inhibition and Behavioral Activation Scale - Activation Fun Seeking Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Behavioral Inhibition and Behavioral Activation Scale- Activation Fun Seeking subscale is a well-validated measure that assesses for trait-like behavioral fun seeking, similar to excitement seeking and surgency on other measures of activation. Participants respond to four items, rated on a 4-point Likert scale (1 - Very true for me to 4 - Very false for me) to indicate their general levels of fun/excitement seeking. Higher scores on the measure indicate higher fun seeking. Total possible scores range from 4 to 16.
Change from baseline on Behavioral Inhibition and Behavioral Activation Scale - Activation Reward Responsiveness Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Behavioral Inhibition and Behavioral Activation Scale- Activation Reward Responsiveness subscale is a well-validated measure that assesses for trait-like behavioral sensitivity to reward. Participants respond to five items, rated on a 4-point Likert scale (1 - Very true for me to 4 - Very false for me) to indicate their general levels of reward sensitivity. Higher scores on the measure indicate higher pleasure from reward and reward seeking. Total possible scores range from 5 to 20.
Change from baseline on Quality of Life Enjoyment and Satisfaction Questionnaire at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Quality of Life Enjoyment and Satisfaction Questionnaire is a measure which assesses current levels participant satisfaction in many domains of their life (e.g., social and romantic relationships, work/school, health, overall wellbeing). Participants respond to sixteen items, rated on a 5-point Likert scale (1 - Very Poor to 6 - Very Good) to indicate their levels of quality of life and life satisfaction during the past week. Higher scores on the measure indicate greater satisfaction. Total possible scores range from 16 to 80.
Change from baseline on Dimensional Anhedonia Rating Scale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Dimensional Anhedonia Rating Scale is a measure which assesses participant current levels of hedonic capacity, or ability to feel pleasure. Participants fill in two experiences that they typically enjoy across four domains (favorite sensory experiences, favorite foods, favorite social activities, favorite pastimes/hobbies) and then rate how much they would enjoy, spend time on, desire for, and interest of each domain, rated on a 5-point Likert scale (1 - Not at All to 5 - Very Much). These ratings are summed to index overall desire for, satisfaction with, and likelihood of pursuing favorite activities at the trait-level (i.e., no specific timeframe). Higher scores indicate greater hedonic capacity. Total possible scores range from 16 to 80.
Change from baseline on Intolerance of Uncertainty Scale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Intolerance of Uncertainty Scale is a measure which assesses trait-like tolerance of uncertainty across numerous life domains. Participants respond to 27 items, rated on a 5-point Likert scale (0 - Not at all characteristic to 4 - Entirely characteristic) to indicate their general tolerance of uncertainty. Higher scores on the measure indicate greater intolerance of uncertainty. Total possible scores range from 0 to 108.
Change from baseline on Multidimensional Psychological Flexibility Inventory (short form) - Flexibility Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Multidimensional Psychological Flexibility Inventory (short form)- Flexibility Subscale is a measure which assesses various aspects of psychological flexibility in line with the hexaflex model of psychological flexibility. Participants respond to twelve items, rated on a 6-point Likert scale (0 - Never true to 5 - Always true) to indicate their level of agreement with each statement regarding facets of flexibility over the past two weeks. Higher scores on the subscale indicate greater flexibility. Total possible scores range from 0 to 60.
Change from baseline on Multidimensional Psychological Flexibility Inventory (short form) - Inflexibility Subscale at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Multidimensional Psychological Flexibility Inventory (short form)- Inflexibility Subscale is a measure which assesses various aspects of psychological inflexibility in line with the hexaflex model of psychological flexibility. Participants respond to twelve items, rated on a 6-point Likert scale (0 - Never true to 5 - Always true) to indicate their level of agreement with each statement regarding facets of inflexibility over the past two weeks. Higher scores on the subscale indicate greater inflexibility. Total possible scores range from 0 to 60.
Change from baseline on Self-Compassion Scale Short Form at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Self-Compassion Scale Short Form is a measure which assesses an individual's general level of self-directed compassion when they are going through difficulties. Participants respond to twelve items, rated on a 5-point Likert scale (1 - Almost Never to 5 - Almost Always) to indicate their level of agreement with each statement regarding how self-compassionate they are with themselves. Higher scores on the scale indicate greater levels of self-compassion. Total possible scores range from 12 to 60.
Change from baseline on Becks Depression Inventory II at two weeks post-intervention | Baseline and Two weeks post-intervention
  The Becks Depression Inventory II is a measure which assesses participant current levels of depression over the past two weeks. Participants respond to 21 items, rated on a 4-point Likert scale (0 - Not at all to 3 - Completely) to indicate how much they feel each symptom of depression. Higher scores on the measure indicate greater depression. Total possible scores range from 0 to 63.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, Ph.D., Principal Investigator — Univeristy of North Carolina Chapel Hill
Locations (1):
- Carolina Center for Neurostimulation, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data (IPD) and supporting information will be available nine to thirty-six months following publication.
Access Criteria: Individual researchers and research groups will be able to request access to deidentified IPD and supporting information with approved IRB, IEC, or REB and an executed Data Use Agreement (DUA) with University of North Carolina (UNC) Chapel Hill.
URL: https://osp.unc.edu/contracting/contracting/